CLINICAL TRIAL: NCT03397758
Title: Non-surgical Treatment for Eye Bag Using AGNES(Radiofrequency Device) With Micro-insulated Needle
Brief Title: Treatment for Eye Bag Using Micro-insulated Needle Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-1512/327-006
Record Dates: First submitted 2017-12-18; First posted 2018-01-12 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2017-12

CONDITIONS: Sagging Eyelid Skin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study population (Experimental): They were treated with AGNES micro-insulated needles with RF applicators in two separate sessions, at intervals of four weeks.
  Interventions: Device: Study population

INTERVENTIONS:
Device: Study population — First, periorbital area was treated with the short needles (exposure time 150ms, power 9W) to tighten the overlying dermis. Then, the fat pocket itself was treated additionally with the long needle (exposure time 400ms, power 9W).
  Other Names: AGNES (needle radiofrequency device)

SUMMARY:
The investigators treated twenty-four subjects with lower eyelid fat bulging using the needle radiofrequency system. After treatment, a three-dimensional photogrammetry system was used to objectively measure the change in height of the fat bulge.

DETAILED DESCRIPTION:
Materials and Methods

Subjects

Twenty-four volunteers (4 males and 20 females) with lower eyelid fat bulging were enrolled in this study. The average age of these subjects was 56±6.28 years. The exclusion criteria were as follows: Prior cosmetic facial surgery within the past 1 year, placement of tissue fillers within the last 6 months, laser therapy or chemical peeling of midface within the preceding 3 months, and the use of topical retinoids for the face within the past 1 month. The study protocol was approved by the institutional review board Seoul National University Bundang Hospital and informed consent was obtained from all subjects prior to participation.

Treatment protocol

All treatments were performed under local anesthesia with 1% lidocaine and 1:100,000 epinephrine. To minimize the impact on the treatment area, the least amount of anesthesia required was injected. The amount of AGNES micro-insulated needles with radiofrequency applicators (Gowoonsesang Cosmetics Co, Seongnam, Gyeonggi, Korea) were used to treat the lesions. This device is a monopolar radiofrequency system with 1MHz wavelength. The needles were composed of two parts: The proximal insulated area and the distal non-insulated area. Proximal insulation preserves the epidermis from thermal damage, allowing the procedure to be non-ablative and minimally-invasive.

Subjects were treated in two separate sessions, at intervals of four weeks. Two types of needle tips were used sequentially in each session; one is a tip with three 1.5mm-length short needles with proximal 0.3mm insulation, while the other is a tip with single 5mm-length long needle with proximal 2.5mm insulation. First, periorbital area was treated with the short needles (exposure time 150ms, power 9W) to tighten the overlying dermis. Then, the fat pocket itself was treated additionally with the long needle (exposure time 400ms, power 9W) to tighten the orbital septum and directly damage the fat cells. Each insertion site was about 1mm apart. After treatment, the treated areas were cooled with ice packs for 20min and topical antibiotic was applied. All subjects were instructed to cleanse their face gently with tap water and avoid sun exposure until next day.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult with age of 40s or more
* Who has lower eyelid fat bulging

Exclusion Criteria:

* History of keloid or hypertrophic scar
* Pregnant woman,
* On breast feeding
* Active skin disease on lesional skin
* Who has severe allergy
* History of bleeding disorder

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
The changes of height of fat bulging | up to 24weeks
  To height of fat bulging was determined as an arbitrary reference plane that links the three points: two points where the right and the left mid pupillary lines meet at each lower eyelid, and the other one point at the pogonion (the most anterior part on the chin). Then, the distance from this reference plane to the highest point of fat bulging was defined as the height of fat bulging.

CONTACTS AND LOCATIONS:
Overall Officials: Chang Hun Huh, MD, PhD, Study Chair — Department of Dermatology, Seoul National University Bundang Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chan NP, Shek SY, Yu CS, Ho SG, Yeung CK, Chan HH. Safety study of transcutaneous focused ultrasound for non-invasive skin tightening in Asians. Lasers Surg Med. 2011 Jul;43(5):366-75. doi: 10.1002/lsm.21070. PMID 21674541
- [Background] Lee JW, Kim BJ, Kim MN, Ahn GY, Aso H. Selective sebaceous gland electrothermolysis as a treatment for acne: a prospective pilot study. Int J Dermatol. 2012 Mar;51(3):339-44. doi: 10.1111/j.1365-4632.2011.05255.x. PMID 22348573
- [Background] Pak CS, Lee YK, Jeong JH, Kim JH, Seo JD, Heo CY. Safety and efficacy of ulthera in the rejuvenation of aging lower eyelids: a pivotal clinical trial. Aesthetic Plast Surg. 2014 Oct;38(5):861-8. doi: 10.1007/s00266-014-0383-6. Epub 2014 Aug 7. PMID 25099495
- [Background] Akita H, Sasaki R, Yokoyama Y, Negishi K, Matsunaga K. The clinical experience and efficacy of bipolar radiofrequency with fractional photothermolysis for aged Asian skin. Exp Dermatol. 2014 Oct;23 Suppl 1:37-42. doi: 10.1111/exd.12391. PMID 25234835
- [Background] Bernardini FP, Cetinkaya A, Devoto MH, Zambelli A. Calcium hydroxyl-apatite (Radiesse) for the correction of periorbital hollows, dark circles, and lower eyelid bags. Ophthalmic Plast Reconstr Surg. 2014 Jan-Feb;30(1):34-9. doi: 10.1097/IOP.0000000000000001. PMID 24398484